CLINICAL TRIAL: NCT00589134
Title: The Effects of Estradiol and Progesterone on Arginine Vasopressin Regulation and Serum Sodium Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Craig Horswill, Gatorade Sports Science Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0508000538
Record Dates: First submitted 2008-01-02; First posted 2008-01-09 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2010-07

CONDITIONS: Exercise Induced Hyponatremia
MeSH Terms: interventions — ganirelix

ARMS (1):
- 1 (Experimental): type of beverage
  Interventions: Dietary Supplement: Gatorade Endurance Formula; Other: ganirelix acetate

INTERVENTIONS:
Dietary Supplement: Gatorade Endurance Formula — carbohydrate electrolyte beverage
Other: ganirelix acetate — GnRH antagonist, subcutaneous injection, 0.25 mg/day for 21 days.
  Other Names: Antagon

SUMMARY:
Women are at greater risk for exercise-induced hyponatremia (low blood sodium concentration) and this risk has been attributed to their lower body weight and size, excess water ingestion and longer racing times relative to men. While these factors contribute to the greater incidence of hyponatremia in women, it is likely that their greater levels of estradiol in plasma and/or tissue also play a role in increasing the risk of hyponatremia in women. More importantly, estradiol may also leave women more susceptible to the extreme consequences of hyponatremia (i.e. brain damage, death). Hyponatremia is generally attributed to inappropriately elevated levels of the hormone arginine vasopressin (AVP). AVP is the most important hormone controlling water retention in the kidney. Earlier studies in our laboratory have demonstrated that estradiol lowers the threshold for thirst sensation and AVP release during exercise. The purpose of these studies is to test the hypotheses that in women with a history of hyponatremia, estradiol lowers the thresholds for thirst and AVP release, leading to greater fluid retention, lower blood sodium concentration during endurance exercise in the heat. However, we further hypothesize that progesterone administration along with estradiol administration will attenuate the effect of estradiol on the regulation of thirst and AVP, normalize fluid retention, and serum sodium concentration during endurance exercise in the heat. In women without a history of hyponatremia, we expect that estradiol administration will lower the thresholds for thirst and AVP release, but will not increase fluid retention or reduce blood sodium concentration during endurance exercise in the heat. We hypothesize that progesterone administration along with estradiol administration will attenuate the effect of estradiol on thirst and AVP, but have no effect on fluid retention or serum sodium concentration during endurance exercise in the heat. To test these hypotheses, women will perform endurance exercise in the heat under three hormonal conditions: 1) during Gonadotropin-releasing hormone (GnRH) antagonist alone--which will suppress estradiol and progesterone; 2) during GnRH antagonist+estradiol; and 3) during GnRH antagonist+estradiol+ progesterone. During exercise, fluid will be replaced with either water or a carbohydrate-electrolyte beverage (random assignment).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (18-35 yrs) with and without previous exercise induced hyponatremia

Exclusion Criteria:

* conditions that would preclude safe exercise or safe use of hormones

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
osmotic regulation of AVP | 3 years

SECONDARY OUTCOMES:
temperature responses | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, PhD, Principal Investigator — John B. Pierce Laboratory
Locations (1):
- John B. Pierce Laboratory, New Haven, Connecticut, United States